CLINICAL TRIAL: NCT01705808
Title: Administration of Protein C Concentrates in Adult Critically Ill Septic Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, Head of Research, Department of Anesthesiology and Intensive Care, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSR/40/04/12
Record Dates: First submitted 2012-07-25; First posted 2012-10-12 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Protein C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Protein C concentrate (Experimental)
  Interventions: Drug: Protein C concentrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Protein C concentrate

INTERVENTIONS:
Drug: Protein C concentrate

SUMMARY:
Severe sepsis and septic shock are life threatening medical emergencies and are among the most significant challenges in critical care. Case reports and case series suggest that plasma-derived protein C concentrate may improve the outcome of patients with acquired protein C deficiency. Evidence has accumulated on the clinical relevance of the PC pathway in modulating overwhelming inflammation and preventing coagulation derangements, two key mediators of organ damage, and thus of mortality and morbidity, in sepsis. The experience collected through these studies shows that PC is safe, in that it is not associated with bleeding or severe allergic complications,and possibly useful, at least to improve the coagulation abnormalities brought about by sepsis. Unfortunately, however, all we know comes from case series or case reports or an underpowered randomized controlled study. A randomized clinical trial, adequately powered for mortality or clinically relevant outcome, is necessary to confirm PC efficacy.The aim of this study is to demonstrate that Protein C zymogen has clinically relevant implications in terms of reduction of thromboembolic events, 30 days mortality, length of intensive care and hospital stay, time on mechanical ventilation, length of ICU and hospital stay. The study will also confirm that there is no bleeding concern with the use of Protein C concentrates.The study drug will be administered in the Intensive Care Unit for 72 hours and the patients observed till ICU discharge. Telephone followup will be performed at 30 days and at one year.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* At least one of the following 3 criteria:

  * venous-venous extra corporeal membrane oxygenation (ECMO) for septic adult respiratory distress syndrome (ARDS)
  * septic disseminated intravascular coagulopathy (DIC)
  * sepsis induced organ dysfunction associated with a clinical assessment of high risk of death

Exclusion Criteria:

* Previous unusual response to PC or any of their components (murine proteins and heparin)
* PC administration or inclusion in other randomized protocols in the previous 30 days
* Do not resuscitate orders
* Refractory cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of number of participant with mortality and/or prolonged ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele di Milano, Italy, Milan, Milano, Italy